CLINICAL TRIAL: NCT04454762
Title: A Phase II Study to Evaluate the Safety, Tolerability and Efficacy of Cabozantinib in Patients With Hepatocellular Carcinoma (HCC) and Impaired Liver Function (Child-Pugh Score B7-8)
Brief Title: A Study to Evaluate the Safety, Tolerability and Efficacy of Cabozantinib in Patients With Hepatocellular Carcinoma and Impaired Liver Function
Acronym: CaboCHILD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Interdisciplinary Center Clinical Trials (IZKS), University Medical Center Mainz (Unknown)
Responsible Party: Principal Investigator, Marcus-Alexander Wörns, Senior consultant, Department of Internal Medicine I, Johannes Gutenberg University Mainz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CaboCHILD
Record Dates: First submitted 2020-06-22; First posted 2020-07-01 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; HCC; Child-Pugh; cabozantinib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (Experimental): 40 mg cabozantinib oral daily. When dose reduction is necessary, it is recommended to reduce to 20 mg daily.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — oral administration (40 mg daily, reduced dose 20 mg daily)
  Other Names: Cabometyx

SUMMARY:
This is an prospective, interventional, non-randomized multicenter phase II study to evaluate the safety, tolerability and efficacy of Cabozantinib as a second-line therapy (after one prior systemic therapy) in patients with intermediate to advanced HCC (BCLC B/C) and concomitant impaired liver function CP score B7-8. Subjects who meet all study eligibility criteria will receive Cabozantinib 40 mg daily orally. Subjects will receive Cabozantinib as long as they continue to experience clinical benefit in the opinion of the Investigator or until there is unacceptable toxicity or the need for subsequent systemic anti-cancer treatment or liver directed local anti-cancer therapy. Treatment may continue in this fashion after radiographic progression as long as the Investigator believes that the subject is still receiving clinical benefit from Cabozantinib and that the potential benefit of continuing Cabozantinib outweighs potential risk. In addition, all subjects will be treated with best supportive care. This excludes systemic anti-cancer therapy and liver-directed local anti-cancer therapy.

ELIGIBILITY:
Main inclusion criteria:

1. Written informed consent
2. Age ≥ 18
3. Histological/cytological or non-invasive (according to EASL/AASLD guidelines) diagnosis of HCC
4. Availability of a recent (up to 28 days old) CT/MRI images of thorax and abdomen
5. Subject's HCC is not amenable to a curative treatment approach (e.g., transplant, surgery, radiofrequency ablation) corresponding to BCLC classification B/C
6. Progression or toxicities following one prior systemic therapy for HCC
7. Recovery to ≤ grade 1 from toxicities related to any prior treatments, unless the adverse events are clinically non-significant and/or stable on supportive therapy
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
9. Adequate hematologic function, based upon meeting the following laboratory criteria within 7 days before enrollment: absolute neutrophil count (ANC) ≥ 1200/mm3 (≥ 1.2 x 109/L); platelets ≥ 60,000/mm3 (≥ 60 x 109/L); hemoglobin ≥ 8 g/dL (≥ 80 g/L)
10. Adequate renal function, based upon meeting the following laboratory criteria within 7 days before enrollment: serum creatinine ≤ 1.5 × upper limit of normal or calculated creatinine clearance ≥ 40 mL/min (using the Cockcroft-Gault equation)
11. Liver function Child-Pugh (CP) score B7-8
12. ALBI (albumin-bilirubin) grade 1-2
13. Alanine aminotransferase (ALT) and aspartate amino-transferase (AST) < 7.0 × upper limit of normal (ULN) within 7 days before enrollment
14. Antiviral therapy per local standard of care if active hepatitis B (HBV) infection
15. Capability to understand and comply with the protocol requirements (e.g. sufficient knowledge of German language to answer the questionnaires, ability to swallow intact tablets).

Main exclusion criteria:

1. Fibrolamellar carcinoma or mixed hepatocellular cholangiocarcinoma
2. Receipt of more than 1 prior systemic therapy for advanced HCC. Additional prior systemic therapies used as adjuvant therapy are allowed.
3. Any type of anti-cancer agent (including investigational) within 2 weeks before enrollment
4. Radiation therapy within 4 weeks (2 weeks for radiation for bone metastases) or radionuclide treatment (e.g., I-131 or Y-90) within 6 weeks of enrollment. Subject cannot be enrolled if there are any clinically relevant ongoing complications from prior radiation therapy.
5. Prior Cabozantinib treatment
6. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 3 months before enrollment. Eligible subjects must be without corticosteroid treatment at the time of enrollment.
7. Concomitant anticoagulation, at therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, low molecular weight heparin (LMWH), thrombin or activated coagulation factor X (FXa) inhibitors, or antiplatelet agents (e.g., clopidogrel). Low-dose aspirin for cardioprotection (per local applicable guidelines), low-dose warfarin (≤ 1 mg/day), and low-dose LMWH are permitted.
8. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

   * Cardiovascular disorders including: Symptomatic congestive heart failure, instable angina pectoris, or serious cardiac arrhythmias, uncontrolled hypertension defined as sustained BP > 150 mm Hg systolic, or > 100 mm Hg diastolic despite optimal antihypertensive treatment, stroke (including TIA), myocardial infarction, or other ischemic event within 6 months before enrollment, thromboembolic event within 3 months before enrollment. Subjects with thromboses of portal/hepatic vasculature attributed to underlying liver disease and/or liver tumor are eligible
   * Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation: tumors invading the GI tract, active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction; abdominal fistula, GI perforation, bowel obstruction, intra-abdominal abscess within 6 months before enrollment, Note: Complete healing of an intra-abdominal abscess must be confirmed prior to enrollment
   * Major surgery within 2 months before enrollment. Complete healing from major surgery must have occurred 1 month before enrollment. Complete healing from minor surgery (e.g., simple excision, tooth extraction) must have occurred at least 7 days before enrollment. Subjects with clinically relevant complications from prior surgery are not eligible
   * Cavitating pulmonary lesion(s) or endobronchial disease
   * Lesion invading a major blood vessel (e.g., pulmonary artery or aorta)
   * Clinically significant bleeding risk within 3 months of enrollment including the following: hematuria, hematemesis, hemoptysis of > 0.5 teaspoon (> 2.5 mL) of red blood, or other signs indicative of pulmonary hemorrhage, or history of other significant bleeding if not due to reversible external factors
   * Other clinically significant disorders such as: Active infection requiring systemic treatment, known infection with human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)-related illness; serious non-healing wound/ulcer/bone fracture; malabsorption syndrome; uncompensated/symptomatic hypothyroidism; requirement for hemodialysis or peritoneal dialysis; history of solid organ transplantation
9. Subjects with untreated or incompletely treated varices with bleeding or high risk for bleeding are excluded with the following clarification: subjects with history of prior variceal bleeding must have been treated with adequate endoscopic therapy without any evidence of recurrent bleeding for at least 6 months prior to study entry and must be stable on optimal medical management (e.g. non-selective beta blocker, proton pump inhibitor) at study entry.
10. Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
11. Women of child-bearing potential (WOCBP) and men who are able to father a child, unwilling to be abstinent or use highly effective methods of birth control that result in a low failure rate of less than 1% per year when used consistently and correctly beginning at informed consent, for the duration of study participation and for at least 4 months after last dose of the study drug. Because oral contraceptives might possibly not be considered as "effective methods of contraception" during the treatment with Cabozantinib, they should be used together with another method, such as a barrier method.
12. Currently receiving any other investigational agent or received an investigational agent within 30 days (or within 5 times the half-life of this agent or its relevant metabolites, the longer period will apply) before the first dose of Cabozantinib.
13. Hepatic encephalopathy Grad I-IV according to CP classification (≥ 2 points) and West Haven Criteria
14. Moderate or severe ascites according to CP classification (≥ 3 points)
15. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 7 days before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) [Safety and Tolerability] | Through study completion, up to approximately 2 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be presented.
Number of Participants Who Discontinue Study Treatment Due to Adverse Events (AEs) [Safety and Tolerability] | Through study completion, up to approximately 2 years
  The number of participants who discontinue study treatment due to an AE will be presented.
ALBI [Safety and Tolerability] | Through study completion, up to approximately 2 years
  Assessment of the Albumin-Bilirubin (ALBI) Grade. Grade range 1-3, with 3 indicating greatest severity
ECOG [Safety and Tolerability] | Through study completion, up to approximately 2 years
  Eastern Cooperative Oncology Group (ECOG) performance status. Score range 0 (normal activity) to 5 (dead).
Child-Pugh [Safety and Tolerability] | Through study completion, up to approximately 2 years
  Used to assess the prognosis of chronic liver disease. Classification of severity of liver disease according to the degree of ascites, total bilirubin and albumin, prothrombin time, and degree of encephalopathy. Each measure is scored 1-3, with 3 indicating greatest severity
Blood pressure [Safety and Tolerability] | Through study completion, up to approximately 2 years.
  mmHg

SECONDARY OUTCOMES:
Overall survival (OS) | Through study completion, up to approximately 2 years
  The time between first application of trial medication to date of death due to any cause.
Progression-free survival (PFS) | Through study completion, up to approximately 2 years
  PFS is defined as the time from first intake of trial medication to the date of the first documentation of progressive disease (PD) or death from any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm.
Objective response rate (ORR) | Through study completion, up to approximately 2 years
  The response rate is defined as the percentage of subjects with a confirmed reduction in tumor size compared to baseline as well as fulfilling the criteria for complete or partial response according to RECIST 1.1.
Pharmacokinetics (PK) of Cabozantinib administration. | 6 weeks
  The plasma concentration of Cabozantinib and possible relevant metabolites will be measured in PK samples.
Health-related quality of life (HRQOL) | Through study completion, up to approximately 2 years
  Assessed by the validated German version of the Chronic Liver Disease Questionnaire (CLDQ-D). The questionnaire contains 29 items which can be grouped into the liver-disease specific domains like activity, fatigue, worries, abdominal symptoms, and systemic symptoms. Each category can be judged separately between the groups. The results of the CLDQ-D score are presented on a 7-point Likert scale. Higher results indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus-Alexander Wörns, Prof. MD, Principal Investigator — University Medical Center Mainz
Locations (1):
- Department of Internal Medicine I, Johannes Gutenberg University Mainz, Mainz, Germany